CLINICAL TRIAL: NCT04607096
Title: Intermittent Fasting to Improve Insulin Secretion
Acronym: IFIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Institute of Human Nutrition (Other); Charite University, Berlin, Germany (Other); University Hospital Carl Gustav Carus (Other); University of Leipzig (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital Heidelberg (Other); University of Luebeck (Other); German Diabetes-Center, Leibniz-Institut in Düsseldorf (Other); German Center for Diabetes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 596/2020BO1
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: PreDiabetes; Diabetes type2; Intermittent Fasting; Insulin Secretion
MeSH Terms: conditions — Prediabetic State; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Participants wil either receive a control diet or join the intermittent fasting group stratified by glycemia (prediabetes/diabetes) as well as by subphenotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prediabetic subjects - cluster 3 (Active Comparator): Presence of a cluster 3 phenotype will be examined according to the parameters described by Wagner et al.(Nat. Med. 2020).
  Interventions: Behavioral: Intermittent fasting; Behavioral: Control diet
- Prediabetic subjects - cluster 5 (Active Comparator): Presence of a cluster 5 phenotype will be examined according to the parameters described by Wagner et al.(Nat. Med. 2020).
  Interventions: Behavioral: Intermittent fasting; Behavioral: Control diet
- Patients with type 2 diabetes - subphenotype: Severe insulin-deficient diabetes (SIDD) (Active Comparator): Presence of a SIDD phenotype will be examined according to the parameters de-scribed Ahlqvist et al. (Lancet Diabetes Endocrinol. 2018 May;6(5):361-369).
  Interventions: Behavioral: Intermittent fasting; Behavioral: Control diet
- Patients with type 2 diabetes - subphenotype: Severe insulin-resistant diabetes (SIRD) (Active Comparator): Presence of a SIRD phenotype will be examined according to the parameters de-scribed Ahlqvist et al (Lancet Diabetes Endocrinol. 2018 May;6(5):361-369).
  Interventions: Behavioral: Intermittent fasting; Behavioral: Control diet

INTERVENTIONS:
Behavioral: Intermittent fasting — The intermittent fasting intervention consists of a decreased daily caloric intake of 400 kcal below individual requirements (Harris Benedict Formula) combined with early time restricted fasting according to the schema 16:8. fasting will be performed over 4 weeks.
Behavioral: Control diet — Control group will be advised to reduce daily caloric intake of 400 kcal below individual requirements (Harris Benedict formula)

SUMMARY:
Type 2 diabetes (T2D) mellitus is a challenge for health care systems as the numbers increases constantly. In 2014, 422 million people had been living with diabetes worldwide. The absolute numbers of people with prediabetes have also grown substantially over 25 years worldwide. In Germany, about 10% of the population has T2D and another 21 % of the population has prediabetes.Overall, 16% of all deaths in Germany are attributable to type 2 diabetes. Macro- and microvascular complications of diabetes imply a significant threat for the patients and are already present in the prediabetic state. Short term and long term complications, the burden of treatment, and reduced quality of life are major burdens of the disease. Accumulating data indicate that currently recommended therapeutic diet regimens in patients with obesity and diabetes are not sustainable on the long term. Novel concepts are therefore urgently needed.

T2D occurs when insulin secretion from pancreatic beta-cells cannot sufficiently be increased to compensate for insulin resistance. Causes of beta-cell dysfunction are heterogeneous. In addition, the most important determinants of diabetes remission are the extend of weight loss and restoration of beta-cell function. In the course of diabetes progression, the inability to recover insulin secretion might identify the state of no return to normal glucose tolerance. It is therefore crucial to improve insulin secretion in treatment and prevention of diabetes. Up to now lifestyle intervention trials in prediabetes or pharmacological intervention trials in diabetes did not show improvement of insulin secretion after intervention. However, one recent small human trial shows that intermittent fasting (early time restricted fasting) is able to improve insulin secretion.Currently, there are no trials that examine the effect of intermittent fasting in individuals with a broad range of impaired glucose metabolism (from prediabetes to diabetes). Recently novel subtypes of diabetes and prediabetes with high risk for the early manifestation of diabetes complications have been identified. Currently, prevention strategies for this high risk individuals have not been examined yet. We will study for the first time the effectiveness of 4 weeks intermittent fasting on changes in insulin secretion capacity in subphenotypes of diabetes and in prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 - 40 kg/m²
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* Subjects with prediabetes (IFG and/or IGT, HbA1c 5,4 % - 6,4 %, subphenotype cluster 3 or 5) or
* Subjects with diabetes mellitus type 2 (diagnosis < 1 year, HbA1c = 6,5 - 9 %, no medical treatment, subphenotype SIDD or SIRD)

Exclusion Criteria:

* Subjects with diabetes mellitus type 1 (GAD-, IA2-AB positive)
* Women during pregnancy and lactation
* Treamtent with any medication effecting on glucose metabolism like anti-diabetic drugs or steroids
* Subjects with a haemoglobin (Hb) ≤ 11.5 g/dl (for males) and Hb ≤ 10.5 g/dl (for females) at screening
* Any pancreatic disease
* Medical history of cancer and/or treatment for cancer within the last 5 years.
* Known current presence or history of severe neurological or psychiatric diseases, schizophrenia, bipolar disorder
* Known history of bariatric surgery
* Severe liver or kidney diseases (Alanine Aminotransferase (ALT [SGPT]), Aspartate Aminotransferase (AST [SGOT]) above 3 x upper limit of normal (ULN) or Glomerular Filtration Rate (eGFR) ≤ 60 ml/min (MDRD formula)
* Systemic infection (CRP > 1 mg/dl)
* Severe diabetic complications like chronic kidney disease (CKD), proliferating retinopathy or symptomatic cardiovascular disease
* Presence of any contraindication for the conduct of an MRI investigation, such as cardiac pacemakers, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators, cochlear implants, insulin pumps and nerve stimulators, prosthetic heart valves etc.
* Persons with limited temperature sensation and / or elevated sensitivity to warming of the body
* Persons with a hearing disorder or a increased sensitivity for loud noises
* Claustrophobia
* Participation in other clinical trials or observation period of competing trials up to 30 days prior to this study
* Refusal to get informed of unexpected detected pathological findings

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in first phase insulin secretion. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effect of intermittent fasting vs. a control diet on glucose stimulated first phase insulin secretion adjusted for insulin sensitivity during an hyperglycemic clamp.

SECONDARY OUTCOMES:
Change in second phase insulin secretion. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effect of intermittent fasting vs. a control diet on glucose stimulated second phase insulin secretion adjusted for insulin sensitivity during an hyperglycemic clamp.
Change in insulin sensitivity. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effect of intermittent fasting vs. a control diet on insulin sensitivity using insulin sensitivity index during an hyperglycemic clamp.
Change in BMI. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effect of intermittent vs. a control diet fasting on BMI.
Change in liver fat content. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting vs. a control diet on liver fat content (%) measured by magnetic resonance spectroscopy (3 T whole body imaging).
Change in pancreatic fat content. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting on pancreatic fat content (%) measured by magnetic resonance spectroscopy (3 T whole body imaging).
Change in body fat content. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting vs. a control diet on total adipose tissue (TAT) measured by magnetic resonance tomography (3 T whole body imaging).
Change in visceral adipose tissue. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting vs. a control diet on visceral adipose tissue (VAT) measured by by magnetic resonance tomography (3 T whole body imaging)
Change in subcutaneous adipose tissue. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting vs. a control diet on subcutaneous adipose tissue (SCAT) measured by by magnetic resonance tomography (3 T whole body imaging)

OTHER OUTCOMES:
Change in brain insulin sensitivity. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting vs. a control diet on brain insulin sensitivity measured by functional magnetic resonance imaging (fMRI) combined with nasal insulin administration.
Change in resting energy expenditure (REE). | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting vs. a control diet on resting energy expenditure measured by indirect calorimetry.
Change in substrate oxidation. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effects of intermittent fasting vs. a control diet on substrate oxidation measured by indirect calorimetry.
Change in proinsulin processing. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effect of intermittent fasting vs. a control diet on first phase proinsulin processing during an hyperglycemic clamp.
Change in glucagon suppression. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effect of intermittent fasting vs. a control diet on glucagon suppression during an hyperglycemic clamp.
Change in insuin clearance. | Before, after 4 weeks and after 24 weeks of lifestyle intervention.
  Effect of intermittent fasting vs. a control diet on insulin clearance during an hyperglycemic clamp.

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - Charité Berlin - Department of Endocrinology and Metabolic Diseases, Berlin
  - Universtiy Hospital Carl Gustav Carus, Dresden
  - German Diabetes Center, Düsseldorf
  - Heidelberg University Hospital - Department of Endocrinology and Metabolism, Heidelberg
  - University Hospital Leipzig - Clinic for Endocrinology and Nephrology, Leipzig
  - University of Luebeck - Institute of Endocrinology and Diabetes, Lübeck
  - Technical University of Munich - Else Kroener-Fresenius-Center for Nutritional Medicine, Munich
  - University Hospital Tuebingen - Institute for Diabetes Research and Metabolic Diseases (IDM), Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heilmann G, Trenkamp S, Moser C, Bombrich M, Schon M, Yurchenko I, Strassburger K, Rodriguez MM, Zaharia OP, Burkart V, Wagner R, Roden M. Precise glucose measurement in sodium fluoride-citrate plasma affects estimates of prevalence in diabetes and prediabetes. Clin Chem Lab Med. 2023 Oct 24;62(4):762-769. doi: 10.1515/cclm-2023-0770. Print 2024 Mar 25. PMID 37870928